CLINICAL TRIAL: NCT01296243
Title: A Phase II Study of Single-agent Tesetaxel in Chemotherapy-naive Patients Who Have Progressive, Castration-resistant Prostate Cancer
Brief Title: Tesetaxel in Chemotherapy-naive Patients With Progressive, Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOP205; PCCTC LOI # c10-071 (Other: Prostate Cancer Clinical Trials Consortium)
Record Dates: First submitted 2011-02-10; First posted 2011-02-15 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Castration-resistant prostate cancer; Tesetaxel; Taxanes; Chemotherapy-naive; Chemotherapy-exposed; Progressive, metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tesetaxel once every 3 weeks (Experimental)
  Interventions: Drug: Tesetaxel

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel capsules will be administered orally once every 21 days until progression, as defined by Prostate Cancer Working Group 2 (PCWG2) criteria. The duration of protocol therapy will not exceed 12 months. Treatment will be initiated at a dose of 27 mg/m2; dose escalation to a maximum of 35 mg/m2 is allowed in Cycle 2 depending on tolerability.
  Other Names: DJ-927

SUMMARY:
Given the activity of docetaxel in patients with progressive, metastatic castration-resistant prostate cancer, this study is being undertaken to evaluate the activity of tesetaxel, an orally bioavailable taxane, in chemotherapy-naive and chemotherapy-exposed patients.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years of age
* Histologically confirmed prostate cancer, currently with progressive disease
* Evidence of metastatic disease
* Castrate level of testosterone (< 50 ng/dL)
* Eastern Cooperative Oncology Group performance status 0 or 1
* Chemotherapy-naïve
* Adequate bone marrow, hepatic, and renal function
* Ability to swallow an oral solid-dosage form of medication

Key Exclusion Criteria:

* History or presence of brain metastasis or leptomeningeal disease
* Operable cancer
* Uncontrolled diarrhea
* Uncontrolled nausea or vomiting
* Known malabsorptive disorder
* Currently active second malignancy other than non-melanoma skin cancers
* Human immunodeficiency virus (HIV) infection based on history of positive serology
* Significant medical disease other than cancer
* Presence of neuropathy > Grade 2 (National Cancer Institute Common Toxicity Criteria [NCI CTC]; v4.0)
* Need for other anticancer treatment
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity
* Less than 2 weeks since use of a medication or ingestion of an agent, beverage, or food that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity
* Less than 4 weeks since use of another investigational agent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-08 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months from the start of treatment

SECONDARY OUTCOMES:
Response rate (RECIST 1.1) among patients with measurable disease | 6 months from the start of treatment
Duration of response among patients with measurable disease | 12 months from the start of treatment
Durable response among patients with measurable disease | 12 months from the start of treatment
Overall survival | 3 years following enrollment of the last subject
Disease-control rate | 6 months from the start of treatment
PSA response rate | Week 12
Progression-free survival | 12 months from the start of treatment
No. (percentage) of subjects with adverse events | Through 30 days after the last dose of tesetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - University of Michigan Health System, Ann Arbor, Michigan
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin